CLINICAL TRIAL: NCT05733338
Title: The Effects of Intermittent Hypoxia on Acute Hypoxic Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Principal Investigator, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IH-AHI
Record Dates: First submitted 2023-01-10; First posted 2023-02-17 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Acute Mountain Sickness
MeSH Terms: conditions — Altitude Sickness

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IH group (Active Comparator): Participants will receive 10 times intermittent hypoxia (oxygen concentration: 13%) intervention before exposure to acute hypoxia environment.
  Interventions: Other: Intermittent Hypoxia
- Control group (Sham Comparator): Participants will receive 10 times sham-hypoxia (oxygen concentration: 21%) intervention in 5 days before exposure to acute hypoxia environment.
  Interventions: Other: Sham Intermittent Hypoxia

INTERVENTIONS:
Other: Intermittent Hypoxia — The intermittent hypoxia protocol refers to four cycles of 10 minutes hypoxia inhaling interval by 5 minutes normoxia, which is performed twice a day (at least 6 hours apart) in 5 days.
  Arms: IH group
Other: Sham Intermittent Hypoxia — The sham intermittent hypoxia protocol refers to 55 minutes normoxia inhaling, which is performed twice a day (at least 6 hours apart) in 5 days.
  Arms: Control group

SUMMARY:
This study intends to further reveal the effectiveness of intermittent hypoxia in preventing acute hypoxic injury.

DETAILED DESCRIPTION:
Acute exposure to hypoxia can induce acute hypoxic injury (AHI), according to the severity of the injury, it can be divided into acute mountain sickness (AMS), high altitude pulmonary edema (HAPE) and high altitude cerebral edema (HACE). AMS is the most common type, it mostly occurs within 6-12 hours after rapidly entering the altitude above 2500m, sometimes within 1h, and can be manifested as headache, nausea, diarrhea, sleep disorders, etc. The incidence of AMS at the altitude of 2500-3000m is 10-20%, which reaches 50-85% at 4500-5000m above sea level.

Intermittent hypoxia (IH) refers to periodic hypoxic-normoxic training performed with brief exposure to hypoxia. Previous studies have found that short-term intermittent hypoxia can increase the sensitivity of hypoxia and reduce the severity of acute hypoxia injury, and alleviate acute hypoxia injury by reducing the inflammatory response caused by hypoxia. Therefore, this study aims to conduct a randomized controlled trial to further reveal the effectiveness of IH and explore its potential mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Informed written consent from the volunteers.
* Healthy volunteers between ages of 18 and 45 years, body mass index (BMI) of 19.0 and 24.9 kg/m2.
* Long-term residence at flatland (altitude of <100 m), not having been to an altitude ≥1500 m in 30 days.
* Resting peripheral oxygen saturation of more than 90%, cerebral oxygen saturation between 58%-82%, heart rate between 60 bpm and 100 bpm, and blood pressure within the normal range (90-130/60-80 mmHg).

Exclusion Criteria:

* History of cardiovascular, cerebrovascular, pulmonary, hepatic, dermatologic, or hematologic diseases.
* History of substance abuse.
* The use of medications or medical devices.
* Pregnancy, hypertension, diabetes mellitus, obesity, sleep apnea and neurological disorders.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute mountain sickness between IH group and control group | After the 6-hour acute hypoxia exposuring.
  A questionnaire called 2018 Lake Louise Scoring System (LLSS) score [0-12] will be used in this primary outcome assessment. The higher LLS scores mean the worse symptoms of acute mountain sickness (AMS).

SECONDARY OUTCOMES:
Concentration of serum parameters between IH group and control group | After the 6-hour acute hypoxia exposuring.
Incidence of intracranial hypertension between IH group and control group | After the 6-hour acute hypoxia exposuring.
  A noninvasive cranial pressure detector will be used to monitor the intracranial pressure.
Incidence of decreased reaction and executive ability between IH group and control group | After the 6-hour acute hypoxia exposuring.
  Related questionnaires will be used to assess the relevant cognitive domain.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No